CLINICAL TRIAL: NCT00294762
Title: A Phase 2 Randomized Study of Tarceva (Erlotinib) as a Single Agent or Intercalated With Combination Chemotherapy in Patients With Newly Diagnosed Advanced Non-small Cell Lung Cancer Who Have Tumors With EGFR Protein Overexpression and/or Increased EGFR Gene Copy Numbers
Brief Title: Erlotinib (Tarceva) as a Single Agent or Intercalated With Combination Chemotherapy in Patients With EGFR Positive NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSI-774-203
Record Dates: First submitted 2006-02-17; First posted 2006-02-22 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; Erlotinib; Tarceva; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib (Experimental): 150 mg erlotinib daily
  Interventions: Drug: Tarceva
- Erlotinib + chemotherapy (intercalated) (Experimental): carboplatin AUC 6 on Day 1 to 21 days, paclitaxel 200 mg/m2 on Day 1 to 21 days, erlotinib 150 mg Days 2-15 for 4 cycles then erlotinib 150 mg daily until progression, withdrawal of consent, or unacceptable toxicity
  Interventions: Drug: Tarceva; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: Tarceva — oral tablet
  Other Names: erlotinib; OSI-774
Drug: carboplatin — IV
  Arms: Erlotinib + chemotherapy (intercalated)
Drug: paclitaxel — IV
  Arms: Erlotinib + chemotherapy (intercalated)

SUMMARY:
This will be the first prospective study where patients will be selected on the basis of two measures of the epidermal growth factor receptor (EGFR) pathway. The study will assess prospectively the efficacy of erlotinib as a single agent or intercalated with chemotherapy in highly selected patients with EGFR overexpression and/or EGFR amplification.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Histologically or cytologically documented non-small cell lung cancer (NSCLC)
* Eastern Cooperative Oncology Group (ECOG)performance status (PS)0, 1, 2
* Radiologically measurable or evaluable disease No prior chemotherapy
* 1 or 2 epithelial growth factor receptor (EGFR) pathway markers positive at screening
* Tumor tissue block or fine needle aspirate

Exclusion Criteria:

* Any concurrent anticancer therapy or radiation
* Other active malignancy
* Uncontrolled brain metastases
* GI abnormalities
* Severe abnormalities of the cornea
* Significant cardiac disease
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (38):
  - Central Hematology Oncology Medical Group Inc., Alhambra, California
  - Comprehensive Blood and Cancer Center(Part of TORI network), Bakersfield, California
  - Bay Area Cancer Research Group, Concord, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA Medical Center, Los Angeles, California
  - North Valley Hematology/Oncology Medical GroupThe Thomas and Dorothy Leavey Cancer Center, Northridge, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Wilshire Oncology Medical GroupThe Robert and Beverly Lewis Family Cancer Care Center, Pomona, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Sansum Santa Barbara Medical Foundation Clinic, Santa Barbara, California
  - Santa Barbara Hematology Oncology Medical Group, Inc., Santa Barbara, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Rocky Mountain Cancer CenterResearch Department, Denver, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - MD Anderson Cancer Ctr - Orlando, Orlando, Florida
  - Gulfcoast Oncology Associates, Tampa, Florida
  - Suburban Hematology-Oncology Associates, Lawrenceville, Georgia
  - Central Georgia Cancer Care, P.C., Macon, Georgia
  - Rush-Presbyterian-St.Luke's Med Ctr, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Norton Healthcare, Inc., Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Univ. of Minnesota Cancer Center, Minneapolis, Minnesota
  - Hematology Oncology Centers of Northern Rockies Research, Billings, Montana
  - Alegent Healthcare, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Hematology-Oncology Associates, SJ, PA - Virtua Health, Mount Holly, New Jersey
  - Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottsville Cancer Clinic, Pottsville, Pennsylvania
  - Boston Baskin Cancer Groupd/b/a U. of Tennessee Cancer Inst., Memphis, Tennessee
  - The West Cancer Clinic, Memphis, Tennessee
  - ACORN, Memphis, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Fletcher Allen Health Care, Burlington, Vermont
  - Cancer Specialists of Tidewater, Ltd., Chesapeake, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - CR UK, Cambridge
  - Peterborough District Hospital, Cambridge
  - Beatson Oncology Centre, Glasgow
  - Mount Vernon Hospital, Middlesex

REFERENCES:
- See also: OSI Pharmaceuticals website — http://www.osip.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was treated 28 March 2006 and the analysis database locked 20 March 2009
Pre-assignment Details: All enrolled patients were randomly assigned to 1 of 2 treatment groups.
Groups:
- Erlotinib + Chemotherapy (Intercalated): carboplatin AUC 6 on Day 1-21 days, paclitaxel 200 mg/m^2 on Day 1-21 days, erlotinib 150 mg Days 2-15 for 4 cycles then erlotinib 150 mg daily until progression, withdrawal of consent, or unacceptable toxicity
Period: Overall Study
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated)
Started | 72 | 71
Completed | 69 | 68
Not Completed | 3 | 3
Not completed — Did not receive study treatment | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated) | Total
Number analyzed (Participants) | 72 | 71 | 143
Age Continuous [Median (Full Range); unit: years] | 63 [31 to 81] | 63 [27 to 90] | 63 [27 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 31 | 75
  Male | 28 | 40 | 68
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 61 | 52 | 113
  Black | 2 | 7 | 9
  Asian | 9 | 4 | 13
  Hispanic | 0 | 8 | 8
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival
Description: Percentage of patients who's disease had not progressed at 6 months. Disease progression defined as radiological and/or symptomatic disease progression or death in absence of progression.
Time Frame: 6 months after first dose
Population: All patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated)
Number analyzed (Participants) | 69 | 68
Percentage of Patients | 30.7 [20.2 to 41.9] | 26.4 [15.9 to 38.0]

2. Secondary Outcome: Progression-free Survival
Description: Median time until disease progression. Disease progression defined as radiological and/or symptomatic disease progression or death in absence of progression.
Time Frame: Until time of disease progression, as assessed every 21 days (maximum 28.8 months)
Population: All patients who received at least 1 dose of study drug
Measure: Median (Full Range); unit: months
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated)
Number analyzed (Participants) | 69 | 68
months | 2.69 [0.03 to 28.85] | 4.57 [0.03 to 24.51]

3. Secondary Outcome: Overall Survival at 12 Months
Description: Percentage of patients alive after 12 months of study treatment
Time Frame: 12 months from 1st dose
Population: All patients who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percent of Patients
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated)
Number analyzed (Participants) | 69 | 68
Percent of Patients | 58.6 [45.6 to 69.5] | 46.4 [33.3 to 58.6]

4. Secondary Outcome: Overall Survival
Description: Median number of months from first study treatment until time of death
Time Frame: From first study treatment until time of death (maximum 29.0 months)
Population: All patients who received at least 1 dose of study drug
Measure: Median (Full Range); unit: Months
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated)
Number analyzed (Participants) | 69 | 68
Months | 16.72 [0.26 to 29.01] | 11.43 [0.49 to 29.04]

5. Secondary Outcome: Best Tumor Response
Description: Change in size of tumor: Complete Response (CR) = no measurable tumor; Partial Response (PR) = 30% decrease in size of measurable tumor; Stable Disease (SD) = measurable tumor size has not changed; Progressive Disease (PD) = measurable tumor larger than at baseline
Time Frame: While receiving study treatment; assessed every 21 days until progression (maximum 28.8 months)
Population: All patients who received at least 1 dose of study drug and who had both a baseline and at least one on-treatment tumor assessment
Measure: Number; unit: Percent of Patients
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated)
Number analyzed (Participants) | 69 | 67
Percent of Patients
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 11.6 | 22.4
  Stable Disease (SD) | 34.8 | 49.3
  Progressive Disease (PD) | 46.4 | 17.9
  Unable to Determine/Not Evaluable | 7.2 | 10.4

6. Secondary Outcome: Duration of Tumor Response
Description: Median length of time that tumor showed any type of response, ie, CR, PR, or SD
Time Frame: While receiving study treatment; assessed every 21 days until progression (maximum 28.8 months).
Population: All patients who had any type of tumor response, ie, CR, PR, or SD
Measure: Median (Full Range); unit: Months
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated)
Number analyzed (Participants) | 32 | 48
Months | 6.4 [1.2 to 26.1] | 4.1 [1.0 to 23.1]

ADVERSE EVENTS:
Time Frame: While on study drug and 30 days after last dose
Description: Adverse events are provided regardless of causality; safety population includes patients who received at least one dose of study drug
Arm/Group | Erlotinib | Erlotinib + Chemotherapy (Intercalated)
Serious Adverse Events (participants affected / at risk) | 27/69 | 27/68
Other Adverse Events (participants affected / at risk) | 67/69 | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=69) | Erlotinib + Chemotherapy (Intercalated) (N=68)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxix (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 2
Cellulitis (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Transient ischaemic attack (Vascular disorders) | 2 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis superfical (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Convulsion (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Spinal chord compression (Nervous system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Heparin-induced thrombocytopenia (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=69) | Erlotinib + Chemotherapy (Intercalated) (N=68)
RASH (Skin and subcutaneous tissue disorders) | 56 | 52 — Pooled skin event terms
Rash (Skin and subcutaneous tissue disorders) | 40 | 34
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 32
Dry skin (Skin and subcutaneous tissue disorders) | 22 | 17
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 10 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 11
Erythema (Skin and subcutaneous tissue disorders) | 9 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 36 | 43
Nausea (Gastrointestinal disorders) | 25 | 42
Constipation (Gastrointestinal disorders) | 13 | 23
Vomiting (Gastrointestinal disorders) | 11 | 25
Dysgeusia (Gastrointestinal disorders) | 8 | 13
Stomatitis (Gastrointestinal disorders) | 9 | 10
Abdominal pain (Gastrointestinal disorders) | 9 | 6
Dry mouth (Gastrointestinal disorders) | 4 | 8
Dyspepsia (Gastrointestinal disorders) | 6 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Oral pain (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 28 | 41
Pyrexia (General disorders) | 4 | 10
Oedema peripheral (General disorders) | 10 | 3
Asthenia (General disorders) | 2 | 9
Chills (General disorders) | 5 | 6
Pain (General disorders) | 4 | 4
Feeling cold (General disorders) | 5 | 2
Chest discomfort (General disorders) | 2 | 3
Influenza like illness (General disorders) | 2 | 3
Mucosal inflammation (General disorders) | 0 | 5
Anorexia (Metabolism and nutrition disorders) | 21 | 31
Dehydration (Metabolism and nutrition disorders) | 2 | 16
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 10
Decreased appetite (Metabolism and nutrition disorders) | 6 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Weight decreased (Investigations) | 15 | 35
Breath sounds abnormal (Investigations) | 3 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 11
Dizziness (Nervous system disorders) | 3 | 10
Headache (Nervous system disorders) | 6 | 4
Hypoaesthesia (Nervous system disorders) | 3 | 4
Neuropathy (Nervous system disorders) | 0 | 6
Paraesthesia (Nervous system disorders) | 4 | 2
Oral candidiasis (Infections and infestations) | 3 | 5
Urinary tract infection (Infections and infestations) | 4 | 4
Rash pustular (Infections and infestations) | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Paronychia (Infections and infestations) | 3 | 2
Insomnia (Psychiatric disorders) | 10 | 18
Depression (Psychiatric disorders) | 7 | 5
Anxiety (Psychiatric disorders) | 5 | 6
Confusional state (Psychiatric disorders) | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 18
Anaemia (Blood and lymphatic system disorders) | 1 | 14
Leukopenia (Blood and lymphatic system disorders) | 2 | 3
Dry eye (Eye disorders) | 4 | 3
Deep vein thrombosis (Vascular disorders) | 6 | 1
Hypotension (Vascular disorders) | 0 | 7
Hot flush (Vascular disorders) | 2 | 3
Tachycardia (Cardiac disorders) | 2 | 3
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less